CLINICAL TRIAL: NCT03749889
Title: Bump to Baby Study
Brief Title: Low Carb vs Normal Carb in Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to provide OBGYN to assist with study for IRB approval
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Kai Ling Kong, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00002745
Record Dates: First submitted 2018-08-28; First posted 2018-11-21 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100 g carbs (Experimental): 100 grams of carbohydrate allowance for the day
  Interventions: Other: 100 g carbs
- MyPlate (Active Comparator): Carbohydrate suggestions based on standard MyPlate. 45-65% kcal intake from carbs.
  Interventions: Other: MyPlate

INTERVENTIONS:
Other: 100 g carbs — Participants will be assigned a diet of 100g carbs max for the day
  Arms: 100 g carbs
Other: MyPlate — 40-65% of daily intake is from carbohydrates
  Arms: MyPlate

SUMMARY:
The overall purpose of this intervention study is to examine whether low-carbohydrate dietary intervention will prevent the development of gestational diabetes mellitus (GDM) in high-risk pregnant women. The results of this study should help further our understanding of how pregnant women can help prevent gestational diabetes mellitus. We hypothesize that a lower carbohydrate diet will prevent the development of GDM.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 years old
* BMI > 30 and/or history of gestational diabetes mellitus
* Currently in first trimester of pregnancy with single fetus (e.g. not twins, triplets, etc.)
* Newborns of current participants

Exclusion Criteria:

* Diabetes (types 1 and 2)
* History of major chronic disease or blood clotting disorders (e.g., cancer, heart disease, kidney disease, hypertension)
* Known fetal anomaly
* History of eating disorders
* Current use of medications that affect appetite or insulin secretion/sensitivity (e.g. stimulants)
* Current use of illegal substances, antipsychotic or opioid substitution medications, alcohol, or tobacco

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 11 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Birth Outcome Questionnaire | 24 months
  Upon delivery of the baby, a birth outcome questionnaire will be collected which includes questions about the delivery and birth of the baby and a question about gestational diabetes. The answer to gestational diabetes or not will be the measure for the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Ling Kong, PhD, Principal Investigator — SUNY Buffalo
Locations (1):
- SUNY Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided